CLINICAL TRIAL: NCT01267279
Title: Effect of Zoledronic Acid on Femoral Bone Loss Following Total Hip Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Spokane Joint Replacement Center (Other)
Responsible Party: Principal Investigator, David F. Scott, MD, PI, Spokane Joint Replacement Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SJRC-Reclast
Record Dates: First submitted 2010-12-24; First posted 2010-12-28 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Zoledronic Acid (Experimental)
  Interventions: Drug: Zoledronic acid

INTERVENTIONS:
Drug: Zoledronic acid — Zoledronic acid per protocol
  Other Names: Reclast
  Arms: Zoledronic Acid
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
In a randomized, double-blind trial, BMD of the operated proximal femur after total hip replacement measured by dual-energy x-ray absorptiometry (DXA) were compared for up to two years in patients receiving IV ZOL 5 mg infusion (n = 27) or placebo (IV saline infusion; n = 24) at two weeks and one year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary elective total hip replacement

Exclusion Criteria:

* Osteoporosis (BMD ≤-2.5)
* Trauma to the operated femur, hip revisions, femoral dysplasia, trochanteric osteotomy, inflammatory arthritis
* Severe renal impairment
* Use of any medications affecting BMD
* Known sensitivity to bisphosphonates
* Severe dental problems, and pregnancy or being able to conceive and not using reliable birth control methods

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2005-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Zoledronic Acid
Started | 24 | 27
Completed | 22 | 21
Not Completed | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Zoledronic Acid | Total
Number analyzed (Participants) | 24 | 27 | 51
Age, Continuous [Mean (Full Range); unit: Years] | 61.8 [51 to 77] | 60.25 [33 to 84] | 61.03 [33 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 11 | 12 | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 24 | 27 | 51

OUTCOME MEASURES:

1. Primary Outcome: Bone Mineral Density (BMD)
Description: Change in bone mineral density (BMD) (per dual energy x-ray absorptiometry (DXA) imaging) from 1 week post-operative data in the Standard and Custom Gruen Zones around the femoral stem.
Time Frame: 2 years post-operative
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | Zoledronic Acid
Number analyzed (Participants) | 22 | 21
Percent change
  Gruen Zone 1: 2 years | -3.97 (15.2) | 14.30 (9.8)
  Gruen Zone 7: 2 years | -27.3 (11.4) | -9.58 (12.4)

ADVERSE EVENTS:
Arm/Group | Placebo | Zoledronic Acid
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/27
Serious Adverse Events (participants affected / at risk) | 2/24 | 3/27
Other Adverse Events (participants affected / at risk) | 0/24 | 2/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=24) | Zoledronic Acid (N=27)
hepatic liver mass (Hepatobiliary disorders) | 1 (1) | 0 (0)
THA revision (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Liver cancer (Hepatobiliary disorders) | 0 (0) | 1 (1)
Muscular atrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=24) | Zoledronic Acid (N=27)
Flu-like symptoms (General disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No